CLINICAL TRIAL: NCT02939300
Title: Phase II Trial of Ipilimumab and Nivolumab in Leptomeningeal Metastases
Brief Title: Ipilimumab and Nivolumab in Leptomeningeal Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Priscilla Brastianos, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-136
Record Dates: First submitted 2016-08-29; First posted 2016-10-20 (Estimated); Results first posted 2022-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Leptomeningeal Carcinomatosis
Keywords: Leptomeningeal Metastases
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination Of Nivolumab with Ipilimumab (Experimental): All patients will be treated based on their primary tumor diagnosis with a combination regimen of Nivolumab and Ipilimumab. Each treatment cycle is 6 weeks; exceptions below.
  * Melanoma:
    * Nivolumab 1 mg/kg and Ipilimumab 3 mg/kg, every 3 weeks for 4 doses.
    * Followed by Nivolumab 480 mg every 4 weeks until disease progression. Each cycle of monotherapy is defined as 8 weeks.
  * Non-small Cell Lung Cancer / Head and Neck Cancer:
    - Nivolumab 3 mg/kg every 2 weeks, and Ipilimumab 1 mg/kg every 6 weeks.
  * Small Cell Lung Cancer / Breast Cancer / Bladder Cancer:
    * Nivolumab 1 mg/kg and Ipilimumab 3 mg/kg, every 3 weeks for 4 doses.
    * Followed by Nivolumab 240 mg every 2 weeks until disease progression.
  * Renal Cell Carcinoma / Other Solid Tumors (not listed above):
    * Nivolumab 3 mg/kg and Ipilimumab 3 mg/kg, every 3 weeks for 4 doses.
    * Followed by Nivolumab 480 mg every 4 weeks until disease progression. Each cycle of monotherapy is defined as 8 weeks.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — * Melanoma:
    - Combination therapy with Nivolumab 1 mg/kg for 4 doses followed by monotherapy Nivolumab 480 mg per cycle.
  * Non-small Cell Lung Cancer / Head and Neck Cancer:
    - Combination therapy with Nivolumab 3 mg/kg
  * Small Cell Lung Cancer / Breast Cancer / Bladder Cancer:
    - Combination therapy with Nivolumab 1 mg/kg for 4 doses followed by monotherapy Nivolumab 240 mg per cycle.
  * Renal Cell Carcinoma / Other Solid Tumors (not listed above):
    * Combination therapy with Nivolumab 3 mg/kg for 4 doses followed by monotherapy Nivolumab 480 mg per cycle.
  Other Names: Opdivo
Drug: Ipilimumab — * Non-small Cell Lung Cancer / Head and Neck Cancer:
    - Combination therapy with Ipilimumab 1 mg/kg
  * Small Cell Lung Cancer / Breast Cancer / Bladder Cancer:
    - Combination therapy with Ipilimumab 3 mg/kg for 4 doses
  * Renal Cell Carcinoma / Other Solid Tumors (not listed above):
    * Combination therapy with Ipilimumab 3 mg/kg for 4 doses
  Other Names: Yervoy

SUMMARY:
This research study is studying a combination of two drugs as a possible treatment for Leptomeningeal Metastases.

The names of the study interventions involved in this study are:

* Ipilimumab
* Nivolumab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial.

Researchers hope to study the effects of the combination of Nivolumab and Ipilimumab. Many cancers use specific pathways, such as programmed death-1 (PD-1), programmed death-ligand-1 (PD-L1), and cytotoxic T lymphocyte antigen-4 (CTLA-4), to evade the body's immune system. Nivolumab and ipilimumab work by blocking the PD-1/PD-L1 and CTLA-4 pathways and thus releasing the brakes on the immune system so it can stop or slow cancer.

The FDA (the U.S. Food and Drug Administration) has approved Nivolumab and Ipilimumab as a treatment option for melanoma, but has not approved them for use when cancer cells spread to the cerebrospinal fluid

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed disease from any solid tumor
* Age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Karnofsky ≥60%)
* Life expectancy of greater than 3 weeks
* Participants must have normal organ and marrow function as defined below, all screening labs should be performed within 10 days of treatment initiation.

Adequate Organ Function Laboratory Values:

Unit key: mcL = microliter, ULN = upper limit normal

* Hematological

  * Absolute neutrophil count (ANC) ≥1500 /mcL
  * Platelets ≥100,000 / mcL
  * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or Erythropoietin (EPO) dependency (within 7 days of assessment)
* Renal
* Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤ Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):

  * Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL
  * Male CrCl = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL
* Hepatic

  * Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
  * Aspartate transaminase (AST) and Alanine transaminase (ALT) ≤ 3 ULN OR ≤ 5 X ULN for subjects with liver metastases
  * Albumin ≥ 2.5 mg/dL
* Coagulation

  * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Creatinine clearance should be calculated per institutional standard.
* Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for Nivolumab to undergo five half-lives) after the last dose of investigational drug.
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of Nivolumab
* Women must not be breastfeeding
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product. Women who are not of childbearing potential, ie, who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception
* Ability to understand and the willingness to sign a written informed consent document.
* Stable dose of dexamethasone 2 mg or less for 7 days prior to initiation of treatment
* Carcinomatous meningitis, as defined by positive cytology

Exclusion Criteria:

* Participants who have had chemotherapy, targeted small molecule therapy or study therapy within 14 days of protocol treatment, or those who have not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 2 weeks earlier. Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Participants who are receiving any other investigational agents.
* Patients should be excluded if they have an active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Subjects are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if > 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of non-autoimmune conditions (eg, delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
* As there is potential for hepatic toxicity with nivolumab or nivolumab/ipilimumab combinations, drugs with a predisposition to hepatoxicity should be used with caution in patients treated with nivolumab-containing regimen.
* Patients should be excluded if they have had prior systemic treatment with an anti-CTLA4 antibody
* Has a known history of active TB (Bacillus Tuberculosis)
* Patients should be excluded if they are positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
* Patients should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). These participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* History of allergy to study drug components
* History of severe hypersensitivity reaction to any monoclonal antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla Brastianos, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts general Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brastianos PK, Strickland MR, Lee EQ, Wang N, Cohen JV, Chukwueke U, Forst DA, Eichler A, Overmoyer B, Lin NU, Chen WY, Bardia A, Juric D, Dagogo-Jack I, White MD, Dietrich J, Nayyar N, Kim AE, Alvarez-Breckenridge C, Mahar M, Mora JL, Nahed BV, Jones PS, Shih HA, Gerstner ER, Giobbie-Hurder A, Carter SL, Oh K, Cahill DP, Sullivan RJ. Phase II study of ipilimumab and nivolumab in leptomeningeal carcinomatosis. Nat Commun. 2021 Oct 12;12(1):5954. doi: 10.1038/s41467-021-25859-y. PMID 34642329

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combination Of Nivolumab with Ipilimumab
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Combination Of Nivolumab With Ipilimumab: All patients will be treated with the combination regimen of Nivolumab at pre-determine dose with Ipilimumab at a pre-determine dose.This will be followed by Nivolumab Monotherapy.
  Each treatment Cycle will last 6 weeks
  Nivolumab
  Ipilimumab
Arm/Group | Combination Of Nivolumab With Ipilimumab
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 54 [36 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 2
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) performance status is a scale used to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis. Scale ranges from 0 to 5 and a lower score indicates a better functional status.
  Participants
    0 = Fully active; no performance restrictions | 4
    1 = Strenuous physical activity restricted; fully ambulatory and able to carry out light work | 10
    2 = Capable of all self-care but unable to carry out work activities.Up and about >50% of waking hrs | 4
Primary tumor diagnosis [Count of Participants; unit: Participants]
  Breast Cancer | 8
  Melanoma | 2
  Anaplastic astrocytoma | 1
  Esophageal adenocarcinoma | 1
  Ependymoma | 1
  Gastroesophageal (GE) junction adenocarcinoma | 1
  Glioblastoma | 1
  Lung adenocarcinoma | 1
  Ovarian | 1
  Small cell lung carcinoma | 1
Brain metastases at the time of leptomeningeal disease (LMD) diagnosis [Count of Participants; unit: Participants]
  Yes | 13
  No | 5
Extracranial disease at the time of leptomeningeal disease (LMD) diagnosis [Count of Participants; unit: Participants]
  Yes | 11
  No | 5
  Unknown | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Survival
Description: Overall Survival (OS) is defined as the time from registration to death due to any cause, or censored at date last known alive.
Time Frame: 3 months
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Of Nivolumab with Ipilimumab
Number analyzed (Participants) | 18
percentage of participants | 44 [24 to 66]

2. Secondary Outcome: Percentage of Participants With Treatment-related Adverse Events
Description: Grade 3 or 4 treatment-related adverse events occurring in at least 15% of participants, based on CTCAE v4.0 criteria.
Time Frame: 2 years
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Of Nivolumab with Ipilimumab
Number analyzed (Participants) | 18
percentage of participants | 33 [16 to 55]

3. Secondary Outcome: Cumulative Incidence of Progressive Disease at 3 Months for Intracranial Sites
Description: Cumulative incidence describes the average probability of developing progressive disease (PD) by immunotherapy response assessment for neuro-oncology (iRANO) criteria. PD is defined as any of the following: (1) >/= 25% increase in 2-dimensional contrast lesions; (2) significant worsened changes on T2-weighted MRI scans; (3) new lesion; or (4) significant clinical decline. Confirmation of progressive disease is based on follow-up imaging for participants without significant clinical decline.
Time Frame: 3 months post-treatment
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Of Nivolumab with Ipilimumab
Number analyzed (Participants) | 18
percentage of participants | 45 [25 to 80]

4. Secondary Outcome: Cumulative Incidence of Progressive Disease at 3 Months for Extracranial Sites
Description: Cumulative incidence describes the average probability of developing progressive disease (PD) by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria. PD is defined as any of the following: (1) >/= 25% increase in 2-dimensional contrast lesions; (2) significant worsened changes on T2-weighted MRI scans; (3) new lesion; or (4) significant clinical decline. Confirmation of progressive disease is based on follow-up imaging for participants without significant clinical decline.
Time Frame: 3 months post-treatment
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Of Nivolumab with Ipilimumab
Number analyzed (Participants) | 18
percentage of participants | 33 [8 to 62]

5. Secondary Outcome: Number of Participants With Leptomeningeal Disease (LMD) Response Post-Treatment
Description: Cerebrospinal fluid (CSF) collection and cytology is done 6-9 weeks after treatment initiation to assess for LMD response, especially complete response or partial response.
  Complete Response is defined as:
  * Reversion to negative CSF cytology (or NA)
  * Disappearance of all disease related symptoms present prior to therapy (or NA)
  * Complete disappearance of all detectable radiographic evidence of disease (or NA).
  Partial Response is defined as:
  * > 50% decrease in malignant CSF cytology
  * Improvement in neurologic symptoms or no worsening of symptoms
  * Improvement in radiographic evidence of disease. No new sites of measurable or assessable central nervous system (CNS) disease.
Time Frame: 6-9 weeks after treatment initiation
Population: Due to the clinical nature of LMD with rapidly progressive disease, the majority participants did not undergo post-treatment lumbar punctures before going off study or passing away. CSF cytology 6-9 weeks after treatment initiation was only obtained on 4 participants, which does not provide statistically meaningful interpretation of data. Individual results are reported below.
Measure: Number; unit: participants
Arm/Group | Combination Of Nivolumab with Ipilimumab
Number analyzed (Participants) | 4
participants
  Complete Response | 0
  Partial Response | 1

6. Secondary Outcome: Extracranial Progression-Free Survival
Description: Extracranial Progression-Free Survival (EPFS) is defined as the time from first dose of study drug to documented extracranial disease progression or death, whichever occurs first. Extracranial disease progression is assessed with CT scans of the chest, abdomen, and pelvis, by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria and immune-related response criteria (irRC) criteria. Progression is defined using RECIST v1.0 as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. The follow-up of participants who have neither died nor progressed at the time of analysis will be censored at the date of last adequate disease assessment.
Time Frame: 2 years
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Combination Of Nivolumab with Ipilimumab
Number analyzed (Participants) | 18
months | 1.94 [1.35 to 4.44]

7. Secondary Outcome: Intracranial Progression-Free Survival
Description: Intracranial Progression-Free Survival (IPFS) is defined as the time from first dose of study drug to documented intracranial disease progression or death, whichever occurs first. Intracranial disease progression is assessed with CT or MRI scans of the brain, using the Response assessment in neuro-oncology (RANO) criteria, which defines progression as:
  * ≥ 25% increase in in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline; or
  * Presence of new lesions; or
  * Worsening of clinical/neurologic status (unless clearly unrelated to the cancer); or
  * Worsening of non-measurable disease.
  The follow-up of participants who have neither died nor progressed at the time of analysis will be censored at the date of last adequate disease assessment.
Time Frame: 2 years
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Combination Of Nivolumab with Ipilimumab
Number analyzed (Participants) | 18
months | 1.93 [1.28 to 2.66]

ADVERSE EVENTS:
Time Frame: 2.5 years
Arm/Group | Combination Of Nivolumab with Ipilimumab
All-Cause Mortality (participants affected / at risk) | 13/18
Serious Adverse Events (participants affected / at risk) | 10/18
Other Adverse Events (participants affected / at risk) | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Of Nivolumab with Ipilimumab (N=18)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (2)
Meningismus (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (2) — Altered mental status
Hypotension (Vascular disorders) | 1 (1) — during surgery
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) — Superior vena cava syndrome
Death NOS (General disorders) | 2 (2)
General disorders and administration site conditions (General disorders) | 2 (2) — Progressive Disease
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Bronchial Compression with RU Collapse
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Of Nivolumab with Ipilimumab (N=18)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (10)
Alkaline phosphatase increased (Investigations) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 4 (8)
Anorexia (Metabolism and nutrition disorders) | 9 (11)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 5 (10)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Blurred vision (Eye disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1) — Eccymosis (Perioribtal, hip, arms, abdomen, ankles)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Chills (General disorders) | 1 (3)
Colitis (Gastrointestinal disorders) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 6 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (6)
Dizziness (Nervous system disorders) | 5 (6)
Dry eye (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dysesthesia (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (7)
Fatigue (General disorders) | 10 (15)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 7 (13)
Gait disturbance (General disorders) | 7 (12)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Headache (Nervous system disorders) | 8 (14)
Hematoma (Vascular disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (4)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infusion related reaction (General disorders) | 1 (1)
INR increased (Investigations) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (4)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lipase increased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Meningismus (Nervous system disorders) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 3 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 6 (9)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Neutrophil count decreased (Investigations) | 2 (3)
Non-cardiac chest pain (General disorders) | 1 (1)
Nystagmus (Nervous system disorders) | 1 (1)
Pain (General disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Platelet count decreased (Investigations) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (7)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Serum amylase increased (Investigations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Somnolence (Nervous system disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 4 (4)
Urinary retention (Renal and urinary disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (7)
Weight gain (Investigations) | 1 (2)
Weight loss (Investigations) | 4 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
White blood cell decreased (Investigations) | 2 (4)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — abdominal fullness
Nervous system disorders - Other, specify (Nervous system disorders) | 2 (3) — Altered Mental Status
Nervous system disorders - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) — aphasia
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — Aspiration Pneumonia (presumed)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Decrease Mobility
Investigations - Other, specify (Investigations) | 1 (1) — Decreased EGFR
Investigations - Other, specify (Investigations) | 1 (1) — Decreased RBC
Eye disorders - Other, specify (Eye disorders) | 3 (3) — Diplopia
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) — Dysuria
Investigations - Other, specify (Investigations) | 2 (2) — Elevated LDH
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Failure to thrive
Herpes simplex reactivation (Infections and infestations) | 1 (1) — genital herpes flare
Hepatitis viral (Infections and infestations) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) — impulsivity
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) — increased thirst
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Intermittent Diaphoresis
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Intraventricular Hemorrhage
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) — Left Elbow Abrasion
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) — Mood Instability
lip pain (Gastrointestinal disorders) | 1 (1) — nerve pain, lower lip
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) — scalp pulsation
Paresthesia (Nervous system disorders) | 3 (3) — legs
Eye disorders - Other, specify (Eye disorders) | 2 (2) — Ptosis
Investigations - Other, specify (Investigations) | 1 (1) — prolonged partial thromboplastin time (PTT) decrease
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) — Right Lower Extremity Hemiparesis
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3 (3) — tachypnea
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) — tongue sensitivity
Investigations - Other, specify (Investigations) | 1 (1) — transaminitis
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) — Worsened Dysmetria
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Shortness of breath, difficulty breathing
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Respiratory Syncytial Virus
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (2) — Muscle soreness
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Neck stiffness
Arm Pain (General disorders) | 2 (2) — Arm pain
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (5)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (4)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) — Thrombocytopenia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT02939300/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT02939300/ICF_001.pdf